CLINICAL TRIAL: NCT00601185
Title: Confocal Reflectance Microscopy of Shave-Biopsy Sites on Skin in Vivo
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-009; NIH R01 EB0027-15,; R44 CA093106-02c; R44CA093106-02 (NIH)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Basal Cell Carcinoma; Melanoma; Squamous Cell Carcinoma; Non-Malignant Skin Disorders
Keywords: 06-009; Confocal reflectance microscopy; shave-biopsy
MeSH Terms: conditions — Carcinoma, Basal Cell; Melanoma; Carcinoma, Squamous Cell | interventions — Microscopy, Confocal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients undergoing a shave biopsy and confocal microscopy.
  Interventions: Procedure: confocal microscopy in vivo

INTERVENTIONS:
Procedure: confocal microscopy in vivo — A dermatologist will perform a shave biopsy according to standard clinical procedures. This study will be carried out after the shave biopsy. The deep surface and the peripheral margins will be imaged on each patient.

SUMMARY:
The purpose of this study is to evaluate a new instrument that shines light and takes digital pictures of skin. The goal is to develop a technique that may enable fast and accurate detection of skin disorders and cancers for future clinical diagnosis and surgical use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing shave-biopsy on an anatomical site that is readily accessible to the VivaScope 1500 (for example, chest, back, legs, arms, cheek, forehead).
* The additional 110 patients for this amendment will be imaged with the newly developed Vivascope 3000 handheld confocal microscope.
* Ability to sign informed consent.
* Age ≥ 18 years.

Exclusion Criteria:

* Shave-biopsy located on a site that is not amenable to confocal imaging (for example, adjacent to the nose, ears or eyes, fingers, toes).
* Inability to give informed consent.
* Known hypersensitivity to adhesive rings.
* Inability to tolerate imaging procedure (i. e., remain relatively still for multiple short durations of 3-4 minutes).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dermatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2006-02-14 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
is to evaluate and quantify the technical feasibility of reflectance CSLM imaging of shave-biopsy sites on skin in vivo. | conclusion of study

SECONDARY OUTCOMES:
To assess the quality of the CSLM images of the biopsy sites to determine a point estimate of the proportion of images that will be of acceptable quality for formal analysis in the planned study of intraoperative margin detection. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kishwer Nehal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center Hauppauge, Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org